CLINICAL TRIAL: NCT00203671
Title: Mycophenolate Mofetil (MMF): A Long-Term Data Evaluation
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Other Study IDs: 04-05-018-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2007-05

CONDITIONS: Kidney Diseases
Keywords: renal; transplant; kidney; rejection; MMF; Mycophenolate Mofetil; outcomes; Kidney Transplantation
MeSH Terms: conditions — Kidney Diseases; Rejection, Psychology

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purposes of this study are:

* To review past clinical use of mycophenolate mofetil (MMF) in kidney transplant patients;
* To discover why doses were modified and how those modifications affected the survival and health of the transplanted kidney; and
* To determine whether, therefore, the side effects of MMF that result in dose alterations are related to outcome.

DETAILED DESCRIPTION:
Objectives:

We propose collecting data on the MMF total daily dose and regimens used in our transplant population from 1995 to 2003. We will assess why doses were modified and how those modifications affected graft survival, and whether, therefore, the side effects of MMF that result in dose alterations are related to outcome.

Implementation

1. Phase I - To describe initial MMF dosing and subsequent changes
2. Phase II - To explore the potential effect of the above on graft outcomes
3. Phase III - To explore reasons for dose changes and how these relate to tolerability

PHASE I

1. The initial maintenance total daily dose of mycophenolate mofetil (MMF, Cellcept) (Frequency distribution of initial maintenance total daily dose in mg/day)

   Include subgroup information about:
   1. Cadaveric donors vs. living donors
   2. Regimen (BID vs. TID vs. QID)
   3. Race (AA vs. Others)
2. Changes in MMF dose from Initial Maintenance Dose (censor patient info at time of rejection or graft loss)

   1. To answer this question we will look at all time points captured within the first post-transplant year, or at 1, 3, 6, 9 and 12 months post-transplant, whichever is fewer.
   2. We will analyze the frequency distribution of daily doses and subgroup by cadaveric donor vs. living donor sub-group.
3. Patients that had no change in MMF total daily dose during their first year post-transplant.

   No dose change is defined as the same MMF dose at all time periods.
4. Patients that had MMF permanently discontinued in their first year post-transplant.
5. Patients that had a dose reduction during their first post-transplant year.
6. Patients that had the frequency of their MMF daily regimen increased (i.e., from BID to TID or QID) during their first post-transplant year.

PHASE II

1. Acute Rejection

   1. Using the data from Statement 2A above we will assess how many patients experienced a treated acute rejection, and stratify by dose into "total-daily-dose groups" as warranted by frequency distribution.
   2. Using the data from Statement 2 B, C, & D above, we will analyze whether MMF discontinuation, dose reduction, or increase in MMF dosing frequency is associated with the incidence of (subsequent) acute rejection?
2. Graft failure

   1. Using the data from Statement 2A above, we will document how many patients had graft failure.
   2. Using the data from Statement 2 B, C, & D above, we will analyze whether MMF discontinuation, MMF dose reduction, or increase in MMF dosing frequency affects the incidence of graft failure?

PHASE III

1. Reasons for Dose Reduction

The side effects that resulted in dose reduction will be documented and the effect of dose reduction in the subsequent period analyzed as above.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients of either a cadaveric or living donor kidney.
* 18 years of age or older.

Exclusion Criteria:

* Multiple organ transplant recipients.
* Prior kidney transplant recipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from existing medical records of 651 UCLA patients who received a kidney transplant, between the dates of January 1, 1995 - December 31st, 2003 All data was reviewed and analyzed as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan H Wilkinson, MD, Principal Investigator — University of California, Los Angeles; Ralph Barbeito, Ph.D., Study Chair — Novartis Pharmaceuticals